CLINICAL TRIAL: NCT07217782
Title: Pain Processing Mechanisms in Patients With Juvenile Arthritis
Brief Title: Pain in Juvenile Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Hadas Nahman-Averbuch, Assistant Professor, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202505170
Record Dates: First submitted 2025-09-19; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JIA (Other): Inclusion:
  1. Age between 9-17
  2. Males and females
  3. English speakers
  4. Able to complete surveys and understand study instructions
  5. Diagnosed or suspected of juvenile arthritis
  Exclusion Criteria
  Participants will not be enrolled if any of the following criteria exist and based on the investigator discretion:
  1. Pregnancy or breastfeeding
  2. (Control Group) Diagnosed with a chronic pain condition
  3. (Control Group) Diagnosed with psychiatric condition including ADHD, anxiety, depression, etc.
  Interventions: Behavioral: Pressure pain thresholds (measured in kilopascal); Behavioral: Cold pain tolerance (duration in seconds)
- Controls (Other): Inclusion:
  1. Age between 9-17
  2. Males and females
  3. English speakers
  4. Able to complete surveys and understand study instructions
  5. Healthy
  Exclusion Criteria
  Participants will not be enrolled if any of the following criteria exist and based on the investigator discretion:
  1. Pregnancy or breastfeeding
  2. (Control Group) Diagnosed with a chronic pain condition
  3. (Control Group) Diagnosed with psychiatric condition including ADHD, anxiety, depression, etc.
  Interventions: Behavioral: Pressure pain thresholds (measured in kilopascal); Behavioral: Cold pain tolerance (duration in seconds)

INTERVENTIONS:
Behavioral: Pressure pain thresholds (measured in kilopascal) — Pressure will be increased continually and participants will be instructed to press a button the first moment they feel pain from the pressure stimulus. The first threshold measurement will be used as a familiarization. The average threshold is calculated from three measurements. Higher value indicates lower experimental pain sensitivity
Behavioral: Cold pain tolerance (duration in seconds) — Cold pain tolerance will be assessed by having participants immerse their hand or foot in a cold (4-12°C) water bath. Tolerance will be defined by the time of hand withdrawal. Pain ratings of cold pain intensity might be obtained periodically, and both pain intensity and pain unpleasantness will be recorded upon hand/foot withdrawal. Higher value indicates lower experimental pain sensitivity

SUMMARY:
Juvenile idiopathic arthritis (JIA) is the most common rheumatologic disease in children. The main symptoms of JIA, which are often the primary focus of treatment, include joint swelling, stiffness, and tenderness. Additional symptoms can include malaise, fatigue, and pain. However, the exact mechanisms contributing to pain are not yet fully understood. Participants will complete a 2.5-hours study session.

In the study session, psychophysical assessments of thermal and pressure stimuli will be performed. In addition, demographic, social, pubertal maturation, and behavioral and psychological factors will be collected via questionnaires. A saliva sample and/or blood draw may occur for the analysis of various immune factors and sex hormones. If a joint aspiration is done as part of their standard of care, we will request a sample of the synovial fluid for analyses of immune, hormonal and/or genetic factors. Participants will have the option to participate in additional optional follow-up study visits (every 3 months, up to 1 year) and to complete monthly surveys asking about their juvenile arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 9-17
2. Males and females
3. English speakers
4. Able to complete surveys and understand study instructions
5. Juvenile arthritis group: diagnosed or suspected of juvenile arthritis
6. Control group: healthy

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. (Control Group) Diagnosed with a chronic pain condition
3. (Control Group) Diagnosed with psychiatric condition including ADHD, anxiety, depression, etc.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Pressure pain thresholds (PPT) (measured in kilopascal) | 1 year
  Differences in PPT between patients and controls.
  Pressure will be increased continually and participants will be instructed to press a button the first moment they feel pain from the pressure stimulus. The first threshold measurement will be used as a familiarization. The average threshold is calculated from three measurements. Higher value indicates lower experimental pain sensitivity
Cold pain tolerance (duration in seconds) | 1 year
  Differences between patients and controls
  Cold pain tolerance will be assessed by having participants immerse their hand or foot in a cold (4-12°C) water bath. Tolerance will be defined by the time of hand withdrawal. Pain ratings of cold pain intensity might be obtained periodically, and both pain intensity and pain unpleasantness will be recorded upon hand/foot withdrawal. Higher value indicates lower experimental pain sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Nahman-Averbuch, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States